CLINICAL TRIAL: NCT02824185
Title: Potential Interest of Combined Fluorocholine Positron Emission Tomography and Magnetic Resonance Imaging (FCH-PET/MRI) for the Selection of Patients Proposed for Curative Treatment of a Hepatocellular Carcinoma
Brief Title: Combined Fluorocholine Positron Emission Tomography and Magnetic Resonance Imaging (FCH-PET/MRI) in Curative Treatment of a Hepatocellular Carcinoma
Acronym: TOMIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL16_0133
Record Dates: First submitted 2016-06-29; First posted 2016-07-06 (Estimated); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Patients Eligible to a Curative Treatment for Primary HCC
Keywords: FCH-PET/MRI; primary HCC; curative treatment; resection; thermo-ablation; transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FCH-PET/MRI (Experimental): FCH-PET/MRI exam performed in addition to the usual examinations for monitoring hepatocellular carcinoma.
  Interventions: Device: PET/MRI system (SIEMENS AG, Munich, Germany; distributed in France by SIEMENS S.A.S, Saint-Denis, France)

INTERVENTIONS:
Device: PET/MRI system (SIEMENS AG, Munich, Germany; distributed in France by SIEMENS S.A.S, Saint-Denis, France) — A PET/MRI examination will be performed once for all included patients, using injected fluorocholine, with a dose of 3MBq/kg, up to 2 months before HCC treatment.

SUMMARY:
Hepatocellular carcinoma (HCC) is the fifth most common cancer in terms of incidence and the second in terms of mortality. At an early stage, which is based on a low number and size of liver nodules and the absence of extra-hepatic locations (Milan criteria), a curative treatment can be performed, i.e. liver transplantation, surgical resection, or thermo-ablation. These treatments can lead to severe complications, so patients benefiting from them must be carefully selected. The correct identification of all HCC lesions at the time of the therapeutic decision is crucial. MRI is the reference examination for diagnosis but its field of exploration is limited to the upper abdominal area and its sensitivity decreases for nodules of less than two centimetres. Such lesions could actually be HCC that will cause early post-operative progression.

Positron Emission Tomography (PET; functional imaging) with fluorodeoxyglucose can provide prognostic information but impacts initial staging in less than 5% of cases. However, PET with fluorocholine (FCH), available in France since 2010, could detect intra- and extra-hepatic HCC lesions not identified by conventional imaging, potentially impacting patient management (e.g. 52% of patients in a small case study).

FCH-PET/MRI could therefore be the ideal examination for the initial staging of HCC, combining in a single multimodality investigation the reference morphological imaging technique and an efficient functional one. The hypothesis of this study is that FCH-PET/MRI is able to detect, in patients eligible for curative treatment, additional preoperative intra- and extra-hepatic early or metastatic HCC unseen or equivocal with conventional imaging (CT and MRI) and responsible for recurrence or disease progression at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Primary HCC proven by histological or imaging examinations (LIRAD 4 or 5)
* Eligible for curative treatment (Barcelona criteria) i.e. hepatic transplantation according to Milan criteria, surgical resection, or thermo-ablation, according to a multidisciplinary decision care committee
* Affiliated to, or a beneficiary of, a social security system
* Written informed consent.

Exclusion Criteria:

* Patient refusing curative treatment
* Patient with HCC not eligible for curative treatment according to conventional imaging (CT, MRI)
* Patient with performance status >1
* Contraindication to MRI
* Pregnant or lactating woman
* Adult ward of court (under guardianship or trusteeship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-06-14 (Actual); Primary Completion 2023-01-02 (Actual); Study Completion 2023-01-02 (Actual)

PRIMARY OUTCOMES:
Specificity of FCH-PET/MRI for the detection of preoperative lesions | 6 months post-treatment
  Specificity of FCH-PET/MRI for the detection of preoperative lesions not visible with conventional imaging techniques and confirmed as being HCC Specificity of preoperative FCH-PET/MRI will be calculated as a ratio of the number of patients with negative FCH-PET/MRI and no additional lesions in histopathology and/or no progressive lesions confirmed at follow-up, to the total number of patients with no additional lesions in histopathology and/or no progressive lesions confirmed at follow-up.

SECONDARY OUTCOMES:
Progression-free survival rates of patients with and without additional lesions visible on FCH-PET/MRI | 24 months post-treatment
Sensitivity of preoperative FCH-PET/MRI for detecting HCC lesions | 6 months post-treatment
  Sensitivity of preoperative FCH-PET/MRI will be determined as a ratio of the number of patients with positive imaging and additional lesions in histopathology and/or progressive lesions confirmed at follow-up, to the total number of patients with additional lesions in histopathology and/or progressive lesions confirmed at follow-up.
Positive and negative predictive value of FCH-PET/MRI | 6 months post-treatment
  Positive predictive value will be calculated from the number of patients with positive imaging and additional lesions in histopathology and/or progressive lesions confirmed at follow-up, and the total number of patients with positive imaging. Negative predictive value will be calculated from the number of patients with negative imaging and no additional lesions in histopathology and/or progressive lesions confirmed at follow-up, and the total number of patients with negative imaging.
Specificity and sensitivity of FCH-PET/MRI compared with preoperative MRI findings for extra-hepatic HCC lesions and for intra-hepatic HCC lesions | FCH-PET/MRI examination, up to 2 months before treatment
FCH-PET/MRI findings (positive or negative, and standardized uptake value ratio between lesions and liver or tissue) compared to HCC differentiation by histopathology | FCH-PET/MRI examination, up to 2 months before treatment
Costs of performing FCH-PET/MRI | FCH-PET/MRI examination, up to 2 months before treatment
  Direct observation of the realization of FCH-PET/MRI, to be able to reconstitute, in the most reliable way, the cost of the examination (micro-costing method).
Incremental cost-effectiveness ratio | 24 months post-treatment
  Modeling of the patient pathway in terms of resource consumption and efficacy, including the completion of FCH-PET/MRI compared to the usual strategy of patient care
Costs avoided and induced by performing FCH-PET/MRI | 24 months post-treatment

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU de Grenoble, Servide d'Hépato-gastro-entérologie, La Tronche
  - HCL, Hôpital Edouard Herriot, service d'hépato-gastro-entérologie, Lyon
  - Hospices Civils de Lyon, Hôpital Edouard Herriot, service d'hépato-gastro-entérologie, Lyon
  - HCL, Hôpital de la Croix-Rousse, service d'Hépato-gastro-entérologie, Lyon